CLINICAL TRIAL: NCT05876962
Title: The Impact of Rapid Diagnostic Methods in the Diagnosis of Fungal Infections in Intensive Care Units of Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara salah abd El mawgoud, Assistant lecturer, Assiut University
Other Study IDs: Diagnosis of fungal infection
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-07

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis of invasive fungal disease remains challenging in the clinical laboratory. The use of matrix-assisted laser desorption/ionization-time of flight mass spectrometry (MALDI-TOF MS) for the identification of filamentous fungi as well as its application for antifungal resistance testing and strain typing Will be evaluated.

DETAILED DESCRIPTION:
Fungal infections are life-threatening opportunistic infections that have emerged as a major cause of morbidity and mortality in critically ill patients. Yeast infections,mainly Candida spp., remain much more frequent than mold infections. Among mold infections, Aspergillus spp. represent the most frequently isolated filamentous fungi in these circumstances .Candida species are the most common cause of nosocomial fungal infections and the fourth most common source of hospital-acquired infections. Candidiasis is an infection caused by Candida, mostly limited to the skin, nails and mucous membranes. However, it can cause serious systemic infections. Candidiasis is an opportunistic infection occurring in presence of predisposing factors like extensive and prolonged administration of broad-spectrum antimicrobials, corticosteroids, immunosuppressive agents and cytotoxic drugs, diabetes mellitus, HIV, chronic renal failure, haemodialysis, renal transplantation or indwelling urinary catheter.The pathogenicity of Candida spp. is related to a combination of microbial factors such as their ability to grow at 37°C, polymorphism, biofilm formation, hydrolytic enzyme secretion, and phenotypic switching. Candida species are identified by different phenotypic methods including examination of their morphological features, analysis of their ability of carbohydrates assimilation and/or fermentation, and their ability of assimilating different nitrogen compounds. Numerous antifungal classes are used to treat Candida infections; polyenes, azoles, echinocandins and allylamines. These antifungals are used with varying efficacy depending on the type, site of infection and the susceptibility of different Candida species. Azoles are the most frequently used antifungal drugs to treat Candida infections as they achieve high success rates even over short durations of therapy. However, resistance among previously susceptible Candida species has emerged following the expanded use of antifungal agents. Antifungal susceptibility testing methods including broth dilution, disk diffusion and E test are now available with species-specific breakpoints developed by The Clinical and Laboratory Standards Institute (CLSI) for multiple antifungal agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all age group and both sex with clinically suspected fungal infection at intensive care units of Assiut university hospital will be included.

Exclusion Criteria:

* -Patients who are on antifungal treatment and refuse to take part will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all age group and both sex with clinically suspected fungal infection at intensive care units of Assiut university hospital will be included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Phenotypically identify percentage of different fungal infections isolated from various clinical specimens in intensive care units. and Assess their antifungal susceptibility pattern. | baseline
  Assess the accuracy of Maldi-TOF in diagnosis of fungal infections

CONTACTS AND LOCATIONS:
Overall Officials: asmaa omar, Study Chair — professor; mohamed zakaria, Study Chair — professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colombo AL, de Almeida Junior JN, Slavin MA, Chen SC, Sorrell TC. Candida and invasive mould diseases in non-neutropenic critically ill patients and patients with haematological cancer. Lancet Infect Dis. 2017 Nov;17(11):e344-e356. doi: 10.1016/S1473-3099(17)30304-3. Epub 2017 Jul 31. PMID 28774702
- [Background] Pappas PG, Lionakis MS, Arendrup MC, Ostrosky-Zeichner L, Kullberg BJ. Invasive candidiasis. Nat Rev Dis Primers. 2018 May 11;4:18026. doi: 10.1038/nrdp.2018.26. PMID 29749387
- [Background] Mayer FL, Wilson D, Hube B. Candida albicans pathogenicity mechanisms. Virulence. 2013 Feb 15;4(2):119-28. doi: 10.4161/viru.22913. Epub 2013 Jan 9. PMID 23302789
- [Background] Neppelenbroek KH, Seo RS, Urban VM, Silva S, Dovigo LN, Jorge JH, Campanha NH. Identification of Candida species in the clinical laboratory: a review of conventional, commercial, and molecular techniques. Oral Dis. 2014 May;20(4):329-44. doi: 10.1111/odi.12123. Epub 2013 May 16. PMID 23679136
- [Background] Vandeputte P, Ferrari S, Coste AT. Antifungal resistance and new strategies to control fungal infections. Int J Microbiol. 2012;2012:713687. doi: 10.1155/2012/713687. Epub 2011 Dec 1. PMID 22187560